CLINICAL TRIAL: NCT01627522
Title: Evaluation of Finastride Effect in Different Dosage on the Amount of Perioperative Bleeding in Transurthral Resection of Prostate
Acronym: TURP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shiraz University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Aminsharifi, Assistant professor of Urology, Shiraz University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 89-01-01-2395
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Benign Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Finastide low dose (Active Comparator): 2 weeks of daily 5mg finastride before operation
  Interventions: Procedure: TURP
- Finastide high dose (Active Comparator): 4 weeks of daily 5mg finastride before operation
  Interventions: Procedure: TURP
- Control (No Intervention): Control

INTERVENTIONS:
Procedure: TURP — Transurthral resection of prostate
  Arms: Finastide high dose; Finastide low dose

SUMMARY:
Preoperative use of finastride will decrease the amount of perioperative blood loss during and after TURP

The effect of finastride on decreasing the amount of perioperative blood loss during and after TURP is dose dependent

Finastride will decrease microvascular density in prostate tissue and this effect is dose dependent

ELIGIBILITY:
Inclusion Criteria:

* Patients with BPH that require TURP

Exclusion Criteria:

* Previous prostate surgery
* Prostate Cancer
* Coagulopathy
* The use of NSAIDs, Anticoagulants, Antiplatelet drugs
* CRF/ESRD

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Perioperative Hb Drop | 24 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faghihi Hospital, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Aminsharifi A, Salehi A, Noorafshan A, Aminsharifi A, Alnajar K. Effect of Preoperative Finasteride on the Volume or Length Density of Prostate Vessels, Intraoperative, Postoperative Blood Loss during and after Monopolar Transurethral Resection of Prostate: A Dose Escalation Randomized Clinical Trial Using Stereolog Methods. Urol J. 2016 Mar 5;13(1):2562-8. PMID 26945662